CLINICAL TRIAL: NCT00317369
Title: A Dose-finding Study of OPC-6535 in Patients With Active Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Efficacy was not cleared at US study
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 197-05-001; JapicCTI-060217
Record Dates: First submitted 2006-04-21; First posted 2006-04-24 (Estimated); Results first posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-01

CONDITIONS: Crohn Disease
Keywords: OPC-6535; Crohn's disease
MeSH Terms: conditions — Crohn Disease | interventions — tetomilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: OPC-6535(Tetomilast)

SUMMARY:
The purpose of this study to examine the safety and efficacy of OPC-6535 and determine its optimal dose by once-daily oral administration at 0, 25, or 50 mg for 8 weeks in combination with a fixed oral dose of 5-aminosalicylic acid (5-ASA) or in combination with a fixed oral dose of 5-ASA and enteral nutrition in patients with active Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active Crohn's disease
* Patients who have a primary lesion in either the small intestine or the large intestine
* Patients who have been receiving an oral 5-ASA formulation at a fixed regimen and at a fixed dose
* Patients who have either never received enteral nutrition or have been receiving enteral nutrition at a fixed intake of 1200 kcal/day or less
* Either inpatient or outpatient

Exclusion Criteria:

* Patients who have an external fistula (including anal fistula) in which persistent drainage is observed (and who require treatment with antibiotics or synthetic antibacterial agents)
* Patients with short bowel syndrome (and who require intravenous nutritional support due to insufficient intestinal nutrient uptake)
* Patients with an artificial anus
* Patients who have a complication of serious infectious disease (intra-abdominal abscess, etc.)
* Patients who have a complication of malignant tumor
* Female patients who are pregnant, lactating, or possibly pregnant, or who wish to become pregnant during the study period

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-05; Primary Completion 2007-07-11 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — Study Director, Division of New Product Evaluation and Development
Locations (8):
- Japan (8):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Touhoku Region

RESULTS

PARTICIPANT FLOW:
Groups:
- OPC-6535 25 mg: 25 mg OPC-6535 orally administered once daily in the morning for 8 weeks.
- OPC-6535 50 mg: 25 mg OPC-6535 orally administered once daily in the morning for the first week, and the dose was increased to 50 mg for the remaining 7 weeks.
- Placebo: 0 mg OPC-6535 orally administered once daily in the morning for 8 weeks.
Period: Overall Study
Arm/Group | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Started | 10 | 9 | 10
Completed | 8 | 7 | 8
Not Completed | 2 | 2 | 2
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OPC-6535 25 mg | OPC-6535 50 mg | Placebo | Total
Number analyzed (Participants) | 10 | 9 | 10 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 10 | 29
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (9.9) | 36.7 (15.0) | 33.4 (6.3) | 35.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 0 | 5
  Male | 6 | 8 | 10 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 10 | 9 | 10 | 29
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 10 | 9 | 10 | 29

OUTCOME MEASURES:

1. Primary Outcome: Clinical Improvement Rate (Number of Subjects Showing Clinical Improvement/Number of Subjects Evaluated x 100) After 8 Weeks of Study Drug Administration
Description: Definition of clinical improvement: Total Crohn's Disease Activity Index (CDAI) score improved by at least 70 points from the baseline score or to below 150 (CDAI < 150: Remission, CDAI > 450: severe disease)
Time Frame: Week 8
Population: Efficacy was evaluated in the subjects who took at least one dose of the study drug and provided postdosing data concerning the efficacy endpoints. Subjects with GCP violations (noncompliance of obtaining informed consent, start of the trial before obtaining informed consent, trial conducted outside the contract period) were to be excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 10 | 9 | 10
percentage of participants | 20.0 [2.5 to 55.6] | 33.3 [7.5 to 70.1] | 10.0 [0.3 to 44.5]

2. Secondary Outcome: Clinical Improvement Rate After 2 and 4 Weeks of Study Drug Administration
Description: Definition of clinical improvement: Total CDAI score improved by at least 70 points from the baseline score or to below 150 (CDAI < 150: Remission, CDAI > 450: severe disease)
Time Frame: Week 2, Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 10 | 9 | 10
percentage of participants
  Week 2 | 20.0 [2.5 to 55.6] | 22.2 [2.8 to 60.0] | 0.0 [0.0 to 30.8]
  Week 4 | 20.0 [2.5 to 55.6] | 22.2 [2.8 to 60.0] | 10.0 [0.3 to 44.5]

3. Secondary Outcome: Remission Rate (Number of Patients Showing Remission/Number of Patients Evaluated x 100) After 2, 4, and 8 Weeks of Study Drug Administration
Description: Definition of remission: Total CDAI score improved to below 150
Time Frame: Week 2, Week 4，Week 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 10 | 9 | 10
percentage of participants
  Week 2 | 10.0 [0.3 to 44.5] | 11.1 [0.3 to 48.2] | 0.0 [0.0 to 30.8]
  Week 4 | 20.0 [2.5 to 55.6] | 11.1 [0.3 to 48.2] | 0.0 [0.0 to 30.8]
  Week 8 | 20.0 [2.5 to 55.6] | 11.1 [0.3 to 48.2] | 0.0 [0.0 to 30.8]

4. Secondary Outcome: Clinical Improvement Rate (50) by Change in Total CDAI Score (Number of Subjects for Each Change/Number of Subjects Evaluated x 100) After 2, 4, and 8 Weeks of Study Drug Administration
Description: Definition of clinical improvement (50) : Total CDAI score improved by at least 50 points from the baseline score or to below 150 (CDAI < 150: Remission, CDAI > 450: severe disease)
Time Frame: Baseline, Weeks 2, 4, and 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 10 | 9 | 10
percentage of participants
  Week 2 | 30.0 [6.7 to 65.2] | 22.2 [2.8 to 60.0] | 10.0 [0.3 to 44.5]
  Week 4 | 30.0 [6.7 to 65.2] | 22.2 [2.8 to 60.0] | 30.0 [6.7 to 65.2]
  Week 8 | 30.0 [6.7 to 65.2] | 33.3 [7.5 to 70.1] | 20.0 [2.5 to 55.6]

5. Secondary Outcome: Mean Change From Baseline in Total CDAI Score After 2, 4, and 8 Weeks of Study Drug Administration
Description: CDAI scores range approximately from 0 to 600, higher scores indicating greater disease activity (CDAI < 150: Remission, CDAI > 450: Very severe). A negative change in mean score indicates improvement.
Time Frame: Baseline, Weeks 2, 4, and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 10 | 9 | 10
score on a scale
  Week 2 | -19.4 (46.5) | -4.1 (57.9) | -8.8 (25.9)
  Week 4 | -17.1 (77.6) | -22.1 (78.2) | -23.5 (32.0)
  Week 8 | -30.3 (60.3) | -32.3 (80.4) | -31.2 (51.4)

6. Secondary Outcome: Mean Change From the Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Score After 8 Weeks of Study Drug Administration
Description: The IBDQ has been frequently adopted in Japanese and overseas clinical assessments as a scale for evaluating the quality of life (QOL) of patients with inflammatory bowel disease. The IBDQ score was calculated as the sum of the responses (each ranging from 1 to 7) to all 32 questions that address symptoms as a result of Crohn's disease: bowel symptoms, systemic symptoms, emotional function, and social function. Total IBDQ score ranges from 32 to 224 with a higher score indicating a better QOL.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 10 | 9 | 10
score on a scale | 11.6 (19.7) | 1.4 (14.6) | 5.0 (17.0)

7. Secondary Outcome: Mean Change From the Baseline in Crohn's Disease Endoscopic Index of Severity (CDEIS) Score After 8 Weeks of Study Drug Administration
Description: Large bowel endoscopic findings were assessed based on the CDEIS. The CDEIS considers deep ulcer, superficial ulcer, lesion ratio of , and ulcer ratio of the 5 pre-defined segments of the colon (small intestine, right colon, transverse colon, left colon, and rectum). The score ranges from 0 to 44 where higher scores indicate more severe disease.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 1
score on a scale |  |  | -4.0

8. Secondary Outcome: Mean Change in C-reactive Protein (CRP) Level From the Baseline After 4 and 8 Weeks of Study Drug Administration
Time Frame: Baseline, Weeks 4 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
Number analyzed (Participants) | 10 | 9 | 10
mg/dL
  Week 4 | -0.65 (0.72) | -1.49 (2.06) | 0.52 (1.19)
  Week 8 | -0.63 (0.99) | -1.21 (1.90) | 1.26 (2.05)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) occurred during the period from treatment initiation to the completion of examinations at Week 8 of the study drug administration, and serious AEs (SAEs) observed prior to the post-trial investigation (from 14 to 21 days after the completion date of the trial period), regardless of the causal relationship with the study drug, were to be reported and analyzed in the trial.
Description: Safety was evaluated in the subjects who took at least one dose of the study drug and provided postdosing data concerning the safety endpoints. Subjects with GCP violations (noncompliance of obtaining informed consent, start of the trial before obtaining informed consent, trial conducted outside the contract period) were to be excluded from the analysis.
Arm/Group | OPC-6535 25 mg | OPC-6535 50 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 2/9 | 0/10
Other Adverse Events (participants affected / at risk) | 9/10 | 9/9 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-6535 25 mg (N=10) | OPC-6535 50 mg (N=9) | Placebo (N=10)
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-6535 25 mg (N=10) | OPC-6535 50 mg (N=9) | Placebo (N=10)
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Anorectal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 4 | 1
Malaise (General disorders) | 2 | 4 | 1
Pyrexia (General disorders) | 0 | 2 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 2
Blood glucose increased (Investigations) | 0 | 2 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0
Glucose urine present (Investigations) | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 2 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Postural dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 4 | 2
Somnolence (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Depressive symptom (Psychiatric disorders) | 0 | 1 | 0
Affect lability (Psychiatric disorders) | 0 | 1 | 0
Residual urine (Renal and urinary disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No